CLINICAL TRIAL: NCT01700712
Title: Acid Production in Dental Plaque After Exposure to Probiotic Bacteria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: BioGaia AB (Industry); Calcin foundation, Denmark (Other)
Responsible Party: Principal Investigator, Mette Kirstine Keller, Reasearch Associate, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-2-2010-112
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Caries
Keywords: Caries, probiotic bacteria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- L. reuteri (DSM 17938 and ATCC PTA 5289; 1x108 CFU (Active Comparator): 2 tablets a day for 2 weeks
  Interventions: Dietary Supplement: Probiotic Lactobacilli reuteri
- Sugar pill (Placebo Comparator): 2 tablets a day for 2 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic Lactobacilli reuteri
  Arms: L. reuteri (DSM 17938 and ATCC PTA 5289; 1x108 CFU
Dietary Supplement: Placebo
  Arms: Sugar pill

SUMMARY:
The increasing interest in probiotic lactobacilli in health maintenance has raised the question of potential risks. One possible side effect could be an increased acidogenicity in dental plaque. The aim of this study was to investigate the effect of probiotic lactobacilli on plaque lactic acid (LA) production in vitro and in vivo.

Methods. subjects (n=18) were given lozenges with probiotic lactobacilli (L. reuteri DSM 17938 and ATCC PTA 5289) or placebo for two weeks in a double-blinded, randomized cross-over trial. The concentration of LA in supragingival plaque samples was determined at baseline and after 2 weeks. Salivary counts of mutans streptococci (MS) and lactobacilli were estimated with chair-side methods.

ELIGIBILITY:
Inclusion Criteria:

* moderate to high counts of salivary mutans streptococci (>104 CFU) as estimated with the Dentocult SM chair-side test,
* no visible open caries lesions or periodontal disease,

Exclusion Criteria:

* smokers,
* ingestion of probiotic bacteria within the last two months,
* ingestion of antibiotics within the last two months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Acid production in plaque after exposure to probiotic bacteria | 2 weeks

SECONDARY OUTCOMES:
Acid producton in plaque after in vitro exposure to probiotic bacteria | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Mette K Keller, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Keller MK, Twetman S. Acid production in dental plaque after exposure to probiotic bacteria. BMC Oral Health. 2012 Oct 24;12:44. doi: 10.1186/1472-6831-12-44. PMID 23092239